CLINICAL TRIAL: NCT01698736
Title: ABO Blood Group Antibody Elimination by a Combination of Semiselective Immunoadsorption Therapy and Membrane Filtration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Principal Investigator, Farsad Eskandary, MD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EK 1540/2012
Record Dates: First submitted 2012-09-26; First posted 2012-10-03 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Immunology
Keywords: ABO isoagglutinins; ABO incompatible transplantation; immunoadsorption; membrane filtration; plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semiselective IA (Active Comparator): Semiselective immunoadsorption (GAM peptide adsorber)
  Interventions: Device: Semiselective IA
- Semiselective IA + membrane filtration (Experimental): Semiselective immunoadsorption (GAM peptide adsorber) in combination with membrane filtration
  Interventions: Device: Membrane filtration; Device: Semiselective IA

INTERVENTIONS:
Device: Membrane filtration — Membrane filtration (Polysulfone)
  Arms: Semiselective IA + membrane filtration
Device: Semiselective IA — Semiselective immunoadsorption (GAM peptide adsorber)

SUMMARY:
* Recipient desensitization protocols were shown to enable successful living donor kidney transplantation across major ABO blood group barriers. For extracorporeal depletion of circulating ABO antibodies plasmapheresis or ABO blood group specific immunoadsorption (IA) are most commonly used.
* The efficiency of semiselective non-antigen specific IA in ABO-incompatible transplantation is currently not well established. One potential drawback of semiselective adsorbers could be an incomplete elimination of IgM.
* This randomized controlled crossover trial was designed to clarify whether membrane filtration, as an adjunct to semiselective IA, can substantially enhance elimination of IgM.

DETAILED DESCRIPTION:
-Background and study aims

ABO-incompatible living donor kidney transplantation offers the possibility to expand the donor pool by approximately 30%. A variety of different desensitization protocols were shown to enable successful transplantation across major ABO barriers. In this context, apheresis for antibody depletion represents the therapeutic mainstay. Two distinct technical principles, plasmapheresis and ABO antigen-specific immunoadsorption, were shown to allow for excellent short- and intermediate-term outcomes. A particular technical advantage of immunoadsorption may be its high selectivity regarding antibody depletion, which precludes major losses of essential plasma constituents, including coagulation factors and albumin, even after treatment of large plasma volumes. Nevertheless, high treatment costs associated with the use of ABO-specific columns (that are not approved for reuse) may limit their widespread clinical application.

The efficiency of semi-selective immunoadsorption technologies regarding ABO antibody depletion and recipient desensitization is less well established. Theoretically, non-antigen-specific immunoglobulin depletion using protein A-, GAM peptide-, or anti-Ig antibody-based adsorbers, could bring about several advantages, such as lower treatment costs associated with the use of reusable twin columns, and the potential to simultaneously deplete antibodies also against HLA antigens. A critical drawback, however, may be an evident inefficiency regarding (ABO-specific) IgM depletion, and this could pose a considerable risk of rejection.

One strategy to overcome the drawback of incomplete IgM depletion could be the use of semiselective immunoadsorption combined with other antibody depletion technologies. In this context, one attractive option could be an enhancement of antibody elimination by connecting a membrane filter (cascade filter) to the immunoadsorption device. We propose to conduct an open randomized crossover study that is designed to see if membrane filtration when applied as an adjunct to semiselective immunoadsorption (GAM peptide adsorbers) is able to enhance anti-ABO IgM elimination to an extent comparable to ABO antigen-specific immunoadsorption. The results of this study, which will enrol 14 patients receiving IA treatment for clinical indications outside the transplantation field, are expected to provide a valuable basis for the use of combined apheresis approaches in the context of ABO-incompatible kidney transplantation.

-Who can participate?

We are planning to recruit 14 adult patients (>18 years, both genders eligible, healthy volunteers not accepted) that are subject to regular routine IA therapy at >1 weekly intervals for clinical indications that are not related to ABO-incompatible transplantation (antibody-mediated autoimmune disorders, such as systemic lupus erythematosus or myasthenia gravis).

-What does the study involve?

For membrane filtration, we will use a membrane filter with documented capacity to eliminate plasma IgM. The study will be conducted in a randomized crossover design (AB vs. BA design; stratified randomization). Treatment consists in IA plus membrane filtration (A) or IA as the sole treatment (B), respectively. The primary study endpoint is the percent reduction of ABO blood group specific IgM. The study is powered to detect a 30% increase in IgM elimination.

-What are the possible benefits and risks of participating?

We do not expect any direct benefits for the study subjects. This pilot study, however, may provide a valuable basis for a future trial evaluating the clinical impact of combined IA plus membrane filtration in ABO incompatible transplantation. Potential risks include: adverse reactions upon exposure to polysulfone (rash, pruritus, fever), reduction in fibrinogen levels and eventually a transient increase in the risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18a
* Blood group A, B or O
* Regular IA treatment for a disease not related to transplantation
* Use of semiselective IA with GAM peptide adsorbers
* IA treatment interval ≥ 7 days

Exclusion Criteria:

* Age ≤ 18a
* Blood group AB (no isoagglutinins)
* No signed consent
* Pregnancy or breast feeding women (exclusion of pregnancy with pregnancy test)
* Severe disease precluding immunoglobulin elimination by IA (e.g. severe infection)
* Elevated risk of bleeding or coagulation disorders that make systemic anticoagulation with heparin impossible
* Hypersensitivity to heparin or HIT
* Hypersensitivity to polysulfone
* Participation in other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Percent reduction in flow cytometric ABO blood group specific IgM serum levels upon a single apheresis treatment | Blood samples will be taken within one hour before (baseline) and within one hour after each apheresis treatment (average apheresis duration 6 hours).

SECONDARY OUTCOMES:
Percent reduction in flow cytometric ABO blood group specific IgG serum levels upon a single apheresis treatment | Blood samples will be taken within one hour before (baseline) and within one hour after each apheresis treatment (average apheresis duration 6 hours).

OTHER OUTCOMES:
Effect on titers of ABO blood group specific IgG (indirect Coombs test) | Blood samples will be taken within one hour before (baseline) and within one hour after each apheresis treatment (average apheresis duration 6 hours).
Effect on titers of ABO blood group specific IgM (direct agglutination test) | Blood samples will be taken within one hour before (baseline) and within one hour after each apheresis treatment (average apheresis duration 6 hours).
Effect on concentrations of total serum IgG | Blood samples will be taken within one hour before (baseline) and within one hour after each apheresis treatment (average apheresis duration 6 hours).
Effect on concentrations of total serum IgM | Blood samples will be taken within one hour before (baseline) and within one hour after each apheresis treatment (average apheresis duration 6 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Georg Böhmig, MD, Principal Investigator — Department of Nephrology, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Wahrmann M, Schiemann M, Marinova L, Kormoczi GF, Derfler K, Fehr T, Stussi G, Bohmig GA. Anti-A/B antibody depletion by semiselective versus ABO blood group-specific immunoadsorption. Nephrol Dial Transplant. 2012 May;27(5):2122-9. doi: 10.1093/ndt/gfr610. Epub 2011 Nov 15. PMID 22086972